CLINICAL TRIAL: NCT01214902
Title: Constraint Induced Movement Therapy (CIMT) in Babies Home Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Prof. Gross- Tsur Varda, SHAARE ZEDEK MEDICAL CENTER
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: chamudotctil
Record Dates: First submitted 2010-07-27; First posted 2010-10-05 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2010-06

CONDITIONS: Hemiplegia; Cerebral Palsy
MeSH Terms: conditions — Hemiplegia; Cerebral Palsy | interventions — Constraint Induced Movement Therapy; Play Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental CIMT (Experimental): Two month home program that includes restricting the non hemiplegic hand an hour a day during play
  Interventions: Device: Constraint induced movement therapy (CIMT)
- Active Play (Active Comparator): Two month home program that includes active use of hemiplegic hand during play one hour a day
  Interventions: Behavioral: play

INTERVENTIONS:
Device: Constraint induced movement therapy (CIMT) — soft mitten worn on the non hemiplegic hand
  Other Names: Modifide constraint induced movoment therapy
  Arms: Experimental CIMT
Behavioral: play — play which encourages the use of the hemiplegic hand
  Arms: Active Play

SUMMARY:
The research objectives are to test the efficacy of a Modified CIMT treatment in babies diagnosed with hemiplegia, treated in a home program, as compared to a control group of babies receiving a parallel home program but with no CIMT.

ELIGIBILITY:
Inclusion Criteria:

* Babies age 7-18 months diagnosed with Hemiplegic cerebral palsy

Exclusion Criteria:

* Epilepsy not treated

Ages: 7 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Assistive Hand Assessment | after two months of treatment
  Evaluation of the use of the hemiplegic hand as an assiting hand in bilateral activities

CONTACTS AND LOCATIONS:
Locations (1):
- ShaareZMC, Jerusalem, Israel

REFERENCES:
- [Derived] Chamudot R, Parush S, Rigbi A, Horovitz R, Gross-Tsur V. Effectiveness of Modified Constraint-Induced Movement Therapy Compared With Bimanual Therapy Home Programs for Infants With Hemiplegia: A Randomized Controlled Trial. Am J Occup Ther. 2018 Nov/Dec;72(6):7206205010p1-7206205010p9. doi: 10.5014/ajot.2018.025981. PMID 30760393
- [Derived] Chamudot R, Parush S, Rigbi A, Gross-Tsur V. Brain Lesions as a Predictor of Therapeutic Outcomes of Hand Function in Infants With Unilateral Cerebral Palsy. J Child Neurol. 2018 Dec;33(14):918-924. doi: 10.1177/0883073818801632. Epub 2018 Oct 11. PMID 30307370